CLINICAL TRIAL: NCT03302299
Title: URBAN ARCH (3/5) Uganda Cohort TB Preventive Therapy for HIV-infected Alcohol Users in Uganda: an Evaluation of Safety Tolerability and Adherence
Brief Title: Alcohol Drinkers' Exposure to Preventive Therapy for TB (ADEPTT)
Acronym: ADEPTT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Boston University (Other); Boston Medical Center (Other); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2U01AA020776-06 (NIH)
Record Dates: First submitted 2017-09-15; First posted 2017-10-05 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Tuberculosis; HIV/AIDS; Alcohol Abuse
Keywords: Adherence; Hepatotoxicity; Phosphatidtylethanol
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; Alcoholism | interventions — Isoniazid; Tablets; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isoniazid & pyridoxine (Experimental): Isoniazid 300 mg oral tablet: 300 mg daily by mouth for 6 months. Pyridoxine 25 mg oral tablet: 25mg daily by mouth for 6 months.
  Interventions: Drug: Isoniazid 300 Mg ORAL TABLET; Drug: Pyridoxine 25 Mg Oral Tablet

INTERVENTIONS:
Drug: Isoniazid 300 Mg ORAL TABLET — The study intervention will include a single arm given (1) 6H: 300 mg INH daily by mouth for 6 months.
  Other Names: INH
Drug: Pyridoxine 25 Mg Oral Tablet — All participants will also receive 25 mg pyridoxine (vitamin B-6) daily by mouth for 6 months for the treatment duration to reduce the risk of INH-induced peripheral neuropathy.
  Other Names: Vitamin B6

SUMMARY:
The Alcohol Drinkers' Exposure to Preventive Therapy for TB (ADEPTT) will examine the safety and tolerability of, and adherence to, 6 months of daily INH (6H) in 300 TB and HIV-infected persons (200 drinkers and 100 non-drinkers) in Uganda. The first aim is to evaluate the safety and tolerability of 6H overall and by level of alcohol use. The second aim is to estimate adherence and compare adherence by level of alcohol use and at 3 and 6 months. Self-reported measures of alcohol use will be augmented by phosphatidylethanol (PEth), an established biomarker of alcohol use. Objective measures of adherence will include electronic pill bottle monitoring and a novel measure of INH exposure, INH concentration in hair. The study will actively monitor for hepatotoxicity using the U.S. standard of care for TB preventive therapy for heavy drinkers and discontinue if any Grade 3/4 toxicities are detected. The investigators will use the safety, tolerability, and adherence results, together with the known efficacy and mortality benefit of TB preventive therapy in HIV-infected persons in SSA, and an established decision analytic model of TB preventive therapy to conduct the third aim: to determine whether the benefits of TB preventive therapy outweigh the toxicity risks for HIV-infected drinkers in resource limited settings. The study will additionally follow the cohort every 6 months after completing INH to monitor drinking and the development of active TB.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the leading cause of mortality in persons with HIV worldwide, accounting for 20-33% of HIV-related deaths, and is a high-priority area of research in HIV/AIDS by the NIH. TB preventive therapy decreases both all-cause mortality and active TB in persons with HIV by 30-50% above and beyond the benefits of antiretroviral therapy (ART) alone. Based on these findings, the World Health Organization (WHO) recommends isoniazid (INH) preventive therapy (IPT) for all persons with HIV in resource constrained settings. However, the WHO warns against the use of IPT in persons with "regular and heavy alcohol use." This exclusion stems from concern for increased hepatotoxicity in heavy drinkers in settings where liver enzymes are not routinely monitored. Heavy drinking in persons with HIV is very common, approximately 25%, in sub-Saharan Africa (SSA). Heavy drinking increases the risk for active TB at least threefold; thus, HIV-infected alcohol users should be prioritized for TB prevention. However, no studies have systematically assessed the safety of TB preventive therapy in heavy drinkers with or without HIV infection. It is critical to examine the safety and tolerability of TB preventive therapy for HIV-infected drinkers, given the high rates of HIV, TB infection, and alcohol comorbidities worldwide. While the risk of toxicity exists, the risk of TB disease could outweigh the toxicity harms. Thus, it is also crucial to determine whether the mortality benefits outweigh the toxicity risks for this significant portion of the HIV-infected population.

In addition, TB preventive therapy is only effective if taken consistently for the full course. Alcohol use is an established risk factor for decreased ART pill taking and active TB treatment discontinuation. Whether HIV-infected drinkers on ART can be adherent to TB preventive therapy is not known. Therefore it is essential to determine the level of adherence to TB preventive therapy by HIV-infected drinkers on ART, thus this study aims to examine adherence to TB preventative therapy as well.

This is a study to examine 6 months of daily INH (6H) among N=300 persons co-infected with HIV and TB. The aims of the study are:

Aim 1: To examine the safety and tolerability of 6H in HIV/TB co-infected drinkers, measured by hepatotoxicity and treatment discontinuation rates. The main aim is to estimate safety and tolerability overall among drinkers (primary) and by level of drinking (secondary).

Aim 2: To determine the level of TB preventive therapy adherence overall among drinkers and by level of drinking, and at 3 and 6 months. The main goal of this aim is to estimate adherence overall among drinkers (primary). Secondarily the investigators will estimate adherence by level of drinking (heavy, current but not heavy drinkers, and non-drinkers) and compare adherence across drinking levels. The investigators hypothesize that adherence will be highest among the non-drinkers.

Aim 3: To determine whether the benefits of providing TB preventive therapy to HIV-infected drinkers in resource-limited settings outweigh the risks compared to no treatment. The investigators hypothesize that providing TB preventive therapy will result in longer life expectancy and quality-adjusted life expectancy than not providing TB preventive therapy (current standard of care).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patient of the MRRH ISS Clinic
3. HIV-infected
4. Consume alcohol (self-reported consumption in the prior 3 months) (2/3) OR prior year non-drinker (1/3)
5. Live within 2 hours of travel time to the ISS Clinic
6. Fluent in either Runyankole or English
7. No ALT/AST elevations (< = 2X ULN) confirmed by testing
8. On ART for at least 6 months
9. No history of active TB, TB treatment, or TB preventive therapy
10. No probable current active TB as determined by symptom screening and followed by chest X-ray and Xpert MTB/RIF (if symptomatic)
11. Positive TST results confirmed by testing

Exclusion Criteria:

1. Plans to move out of the catchment area within 6 months
2. Probable TB via symptom screen and subsequent assessments
3. History or current or past active TB, TB treatment, or TB preventive therapy
4. ALT or AST >2x ULN
5. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Hahn, PhD, MA, Principal Investigator — University of California, San Francisco
Locations (1):
- Mbarara University of Science and Technology/Mbarara Regional Referral Hospital, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No
The investigators will make de-identified data available to investigators with relevant and well-articulated research plans, after the main study analyses have been conducted. No personal identifiers will be shared, and nor identifiers that could be linked back to the original study ID. In addition, some journals require de-identified data to be posted for public access.

REFERENCES:
- [Background] Akolo C, Adetifa I, Shepperd S, Volmink J. Treatment of latent tuberculosis infection in HIV infected persons. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD000171. doi: 10.1002/14651858.CD000171.pub3. PMID 20091503
- [Background] Edessa D, Likisa J. A Description of Mortality Associated with IPT plus ART Compared to ART Alone among HIV-Infected Individuals in Addis Ababa, Ethiopia: A Cohort Study. PLoS One. 2015 Sep 8;10(9):e0137492. doi: 10.1371/journal.pone.0137492. eCollection 2015. PMID 26348618
- [Background] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Background] Ayele HT, Mourik MS, Debray TP, Bonten MJ. Isoniazid Prophylactic Therapy for the Prevention of Tuberculosis in HIV Infected Adults: A Systematic Review and Meta-Analysis of Randomized Trials. PLoS One. 2015 Nov 9;10(11):e0142290. doi: 10.1371/journal.pone.0142290. eCollection 2015. PMID 26551023
- [Background] Golub JE, Pronyk P, Mohapi L, Thsabangu N, Moshabela M, Struthers H, Gray GE, McIntyre JA, Chaisson RE, Martinson NA. Isoniazid preventive therapy, HAART and tuberculosis risk in HIV-infected adults in South Africa: a prospective cohort. AIDS. 2009 Mar 13;23(5):631-6. doi: 10.1097/QAD.0b013e328327964f. PMID 19525621
- [Background] Akolo C, Bada F, Okpokoro E, Nwanne O, Iziduh S, Usoroh E, Ali T, Ibeziako V, Oladimeji O, Odo M. Debunking the myths perpetuating low implementation of isoniazid preventive therapy amongst human immunodeficiency virus-infected persons. World J Virol. 2015 May 12;4(2):105-12. doi: 10.5501/wjv.v4.i2.105. PMID 25964875
- [Background] Rangaka MX, Cavalcante SC, Marais BJ, Thim S, Martinson NA, Swaminathan S, Chaisson RE. Controlling the seedbeds of tuberculosis: diagnosis and treatment of tuberculosis infection. Lancet. 2015 Dec 5;386(10010):2344-53. doi: 10.1016/S0140-6736(15)00323-2. Epub 2015 Oct 26. PMID 26515679
- [Background] Kader R, Govender R, Seedat S, Koch JR, Parry C. Understanding the Impact of Hazardous and Harmful Use of Alcohol and/or Other Drugs on ARV Adherence and Disease Progression. PLoS One. 2015 May 1;10(5):e0125088. doi: 10.1371/journal.pone.0125088. eCollection 2015. PMID 25933422
- [Background] Wandera B, Tumwesigye NM, Nankabirwa JI, Kambugu AD, Parkes-Ratanshi R, Mafigiri DK, Kapiga S, Sethi AK. Alcohol Consumption among HIV-Infected Persons in a Large Urban HIV Clinic in Kampala Uganda: A Constellation of Harmful Behaviors. PLoS One. 2015 May 11;10(5):e0126236. doi: 10.1371/journal.pone.0126236. eCollection 2015. PMID 25962171
- [Background] Kader R, Seedat S, Govender R, Koch JR, Parry CD. Hazardous and harmful use of alcohol and/or other drugs and health status among South African patients attending HIV clinics. AIDS Behav. 2014 Mar;18(3):525-34. doi: 10.1007/s10461-013-0587-9. PMID 23921585
- [Background] Kekwaletswe CT, Morojele NK. Alcohol use, antiretroviral therapy adherence, and preferences regarding an alcohol-focused adherence intervention in patients with human immunodeficiency virus. Patient Prefer Adherence. 2014 Mar 31;8:401-13. doi: 10.2147/PPA.S55547. eCollection 2014. PMID 24729688
- [Background] Medley A, Seth P, Pathak S, Howard AA, DeLuca N, Matiko E, Mwinyi A, Katuta F, Sheriff M, Makyao N, Wanjiku L, Ngare C, Bachanas P. Alcohol use and its association with HIV risk behaviors among a cohort of patients attending HIV clinical care in Tanzania, Kenya, and Namibia. AIDS Care. 2014;26(10):1288-97. doi: 10.1080/09540121.2014.911809. Epub 2014 Apr 29. PMID 24773163
- [Background] Soboka M, Tesfaye M, Feyissa GT, Hanlon C. Alcohol use disorders and associated factors among people living with HIV who are attending services in south west Ethiopia. BMC Res Notes. 2014 Nov 24;7:828. doi: 10.1186/1756-0500-7-828. PMID 25417542
- [Background] Narasimhan P, Wood J, Macintyre CR, Mathai D. Risk factors for tuberculosis. Pulm Med. 2013;2013:828939. doi: 10.1155/2013/828939. Epub 2013 Feb 12. PMID 23476764
- [Background] Lonnroth K, Williams BG, Stadlin S, Jaramillo E, Dye C. Alcohol use as a risk factor for tuberculosis - a systematic review. BMC Public Health. 2008 Aug 14;8:289. doi: 10.1186/1471-2458-8-289. PMID 18702821
- [Background] Rehm J, Samokhvalov AV, Neuman MG, Room R, Parry C, Lonnroth K, Patra J, Poznyak V, Popova S. The association between alcohol use, alcohol use disorders and tuberculosis (TB). A systematic review. BMC Public Health. 2009 Dec 5;9:450. doi: 10.1186/1471-2458-9-450. PMID 19961618
- [Background] Menzies D, Al Jahdali H, Al Otaibi B. Recent developments in treatment of latent tuberculosis infection. Indian J Med Res. 2011 Mar;133(3):257-66. PMID 21441678
- [Background] Hendershot CS, Stoner SA, Pantalone DW, Simoni JM. Alcohol use and antiretroviral adherence: review and meta-analysis. J Acquir Immune Defic Syndr. 2009 Oct 1;52(2):180-202. doi: 10.1097/QAI.0b013e3181b18b6e. PMID 19668086
- [Background] Kendall EA, Theron D, Franke MF, van Helden P, Victor TC, Murray MB, Warren RM, Jacobson KR. Alcohol, hospital discharge, and socioeconomic risk factors for default from multidrug resistant tuberculosis treatment in rural South Africa: a retrospective cohort study. PLoS One. 2013 Dec 13;8(12):e83480. doi: 10.1371/journal.pone.0083480. eCollection 2013. PMID 24349518
- [Background] Sharma SK, Sharma A, Kadhiravan T, Tharyan P. Rifamycins (rifampicin, rifabutin and rifapentine) compared to isoniazid for preventing tuberculosis in HIV-negative people at risk of active TB. Evid Based Child Health. 2014 Mar;9(1):169-294. doi: 10.1002/ebch.1962. PMID 25404581
- [Background] Martinson NA, Barnes GL, Moulton LH, Msandiwa R, Hausler H, Ram M, McIntyre JA, Gray GE, Chaisson RE. New regimens to prevent tuberculosis in adults with HIV infection. N Engl J Med. 2011 Jul 7;365(1):11-20. doi: 10.1056/NEJMoa1005136. PMID 21732833
- [Background] Bliven-Sizemore EE, Sterling TR, Shang N, Benator D, Schwartzman K, Reves R, Drobeniuc J, Bock N, Villarino ME; TB Trials Consortium. Three months of weekly rifapentine plus isoniazid is less hepatotoxic than nine months of daily isoniazid for LTBI. Int J Tuberc Lung Dis. 2015 Sep;19(9):1039-44, i-v. doi: 10.5588/ijtld.14.0829. PMID 26260821
- [Background] Person AK, Sterling TR. Treatment of latent tuberculosis infection in HIV: shorter or longer? Curr HIV/AIDS Rep. 2012 Sep;9(3):259-66. doi: 10.1007/s11904-012-0120-1. PMID 22581360
- [Background] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Background] Ena J, Valls V. Short-course therapy with rifampin plus isoniazid, compared with standard therapy with isoniazid, for latent tuberculosis infection: a meta-analysis. Clin Infect Dis. 2005 Mar 1;40(5):670-6. doi: 10.1086/427802. Epub 2005 Feb 1. PMID 15714411
- [Background] Hahn JA, Dobkin LM, Mayanja B, Emenyonu NI, Kigozi IM, Shiboski S, Bangsberg DR, Gnann H, Weinmann W, Wurst FM. Phosphatidylethanol (PEth) as a biomarker of alcohol consumption in HIV-positive patients in sub-Saharan Africa. Alcohol Clin Exp Res. 2012 May;36(5):854-62. doi: 10.1111/j.1530-0277.2011.01669.x. Epub 2011 Dec 7. PMID 22150449
- [Background] Mave V, Chandanwale A, Kinikar A, Khadse S, Kagal A, Gupte N, Suryavanshi N, Nimkar S, Koli H, Khwaja S, Bharadwaj R, Joshi S, Horng H, Benet LZ, Ramachandran G, Dooley KE, Gupta A, Gandhi M. Isoniazid hair concentrations in children with tuberculosis: a proof of concept study. Int J Tuberc Lung Dis. 2016 Jun;20(6):844-7. doi: 10.5588/ijtld.15.0882. PMID 27155191
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Baliunas D, Rehm J, Irving H, Shuper P. Alcohol consumption and risk of incident human immunodeficiency virus infection: a meta-analysis. Int J Public Health. 2010 Jun;55(3):159-66. doi: 10.1007/s00038-009-0095-x. Epub 2009 Dec 1. PMID 19949966
- [Background] Shuper PA, Neuman M, Kanteres F, Baliunas D, Joharchi N, Rehm J. Causal considerations on alcohol and HIV/AIDS--a systematic review. Alcohol Alcohol. 2010 Mar-Apr;45(2):159-66. doi: 10.1093/alcalc/agp091. Epub 2010 Jan 8. PMID 20061510
- [Background] Amoakwa K, Martinson NA, Moulton LH, Barnes GL, Msandiwa R, Chaisson RE. Risk factors for developing active tuberculosis after the treatment of latent tuberculosis in adults infected with human immunodeficiency virus. Open Forum Infect Dis. 2015 Jan 20;2(1):ofu120. doi: 10.1093/ofid/ofu120. eCollection 2015 Jan. PMID 26034751
- [Background] Volkmann T, Moonan PK, Miramontes R, Oeltmann JE. Tuberculosis and excess alcohol use in the United States, 1997-2012. Int J Tuberc Lung Dis. 2015 Jan;19(1):111-9. doi: 10.5588/ijtld.14.0516. PMID 25519800
- [Background] Shayo GA, Moshiro C, Aboud S, Bakari M, Mugusi FM. Acceptability and adherence to Isoniazid preventive therapy in HIV-infected patients clinically screened for latent tuberculosis in Dar es Salaam, Tanzania. BMC Infect Dis. 2015 Aug 26;15:368. doi: 10.1186/s12879-015-1085-7. PMID 26306511
- [Background] Mosimaneotsile B, Mathoma A, Chengeta B, Nyirenda S, Agizew TB, Tedla Z, Motsamai OI, Kilmarx PH, Wells CD, Samandari T. Isoniazid tuberculosis preventive therapy in HIV-infected adults accessing antiretroviral therapy: a Botswana Experience, 2004-2006. J Acquir Immune Defic Syndr. 2010 May 1;54(1):71-7. doi: 10.1097/QAI.0b013e3181c3cbf0. PMID 19934764
- [Background] Saukkonen JJ, Cohn DL, Jasmer RM, Schenker S, Jereb JA, Nolan CM, Peloquin CA, Gordin FM, Nunes D, Strader DB, Bernardo J, Venkataramanan R, Sterling TR; ATS (American Thoracic Society) Hepatotoxicity of Antituberculosis Therapy Subcommittee. An official ATS statement: hepatotoxicity of antituberculosis therapy. Am J Respir Crit Care Med. 2006 Oct 15;174(8):935-52. doi: 10.1164/rccm.200510-1666ST. PMID 17021358
- [Background] Comstock GW. Prevention of tuberculosis among tuberculin reactors: maximizing benefits, minimizing risks. JAMA. 1986 Nov 21;256(19):2729-30. No abstract available. PMID 3773185
- [Background] Fountain FF, Tolley E, Chrisman CR, Self TH. Isoniazid hepatotoxicity associated with treatment of latent tuberculosis infection: a 7-year evaluation from a public health tuberculosis clinic. Chest. 2005 Jul;128(1):116-23. doi: 10.1378/chest.128.1.116. PMID 16002924
- [Background] LoBue PA, Moser KS. Use of isoniazid for latent tuberculosis infection in a public health clinic. Am J Respir Crit Care Med. 2003 Aug 15;168(4):443-7. doi: 10.1164/rccm.200303-390OC. Epub 2003 May 13. PMID 12746255
- [Background] Tedla Z, Nyirenda S, Peeler C, Agizew T, Sibanda T, Motsamai O, Vernon A, Wells CD, Samandari T. Isoniazid-associated hepatitis and antiretroviral drugs during tuberculosis prophylaxis in hiv-infected adults in Botswana. Am J Respir Crit Care Med. 2010 Jul 15;182(2):278-85. doi: 10.1164/rccm.200911-1783OC. Epub 2010 Apr 8. PMID 20378730
- [Background] Tedla Z, Nguyen ML, Sibanda T, Nyirenda S, Agizew TB, Girde S, Rose CE, Samandari T. Isoniazid-associated hepatitis in adults infected with HIV receiving 36 months of isoniazid prophylaxis in Botswana. Chest. 2015 May;147(5):1376-1384. doi: 10.1378/chest.14-0215. PMID 25340318
- [Background] Menzies D, Long R, Trajman A, Dion MJ, Yang J, Al Jahdali H, Memish Z, Khan K, Gardam M, Hoeppner V, Benedetti A, Schwartzman K. Adverse events with 4 months of rifampin therapy or 9 months of isoniazid therapy for latent tuberculosis infection: a randomized trial. Ann Intern Med. 2008 Nov 18;149(10):689-97. doi: 10.7326/0003-4819-149-10-200811180-00003. PMID 19017587
- [Background] Getahun H, Chaisson RE, Raviglione M. Latent Mycobacterium tuberculosis Infection. N Engl J Med. 2015 Sep 17;373(12):1179-80. doi: 10.1056/NEJMc1508223. No abstract available. PMID 26376149
- [Background] Parsons JT, Rosof E, Mustanski B. The temporal relationship between alcohol consumption and HIV-medication adherence: a multilevel model of direct and moderating effects. Health Psychol. 2008 Sep;27(5):628-37. doi: 10.1037/a0012664. PMID 18823189
- [Background] Braithwaite RS, McGinnis KA, Conigliaro J, Maisto SA, Crystal S, Day N, Cook RL, Gordon A, Bridges MW, Seiler JF, Justice AC. A temporal and dose-response association between alcohol consumption and medication adherence among veterans in care. Alcohol Clin Exp Res. 2005 Jul;29(7):1190-7. doi: 10.1097/01.alc.0000171937.87731.28. PMID 16046874
- [Background] Duraisamy K, Mrithyunjayan S, Ghosh S, Nair SA, Balakrishnan S, Subramoniapillai J, Oeltmann JE, Moonan PK, Kumar AM. Does Alcohol consumption during multidrug-resistant tuberculosis treatment affect outcome?. A population-based study in Kerala, India. Ann Am Thorac Soc. 2014 Jun;11(5):712-8. doi: 10.1513/AnnalsATS.201312-447OC. PMID 24735096
- [Background] Namuwenge PM, Mukonzo JK, Kiwanuka N, Wanyenze R, Byaruhanga R, Bissell K, Zachariah R. Loss to follow up from isoniazid preventive therapy among adults attending HIV voluntary counseling and testing sites in Uganda. Trans R Soc Trop Med Hyg. 2012 Feb;106(2):84-9. doi: 10.1016/j.trstmh.2011.10.015. Epub 2011 Dec 10. PMID 22154974
- [Background] Munseri PJ, Talbot EA, Mtei L, Fordham von Reyn C. Completion of isoniazid preventive therapy among HIV-infected patients in Tanzania. Int J Tuberc Lung Dis. 2008 Sep;12(9):1037-41. PMID 18713501
- [Background] Durovni B, Cavalcante SC, Saraceni V, Vellozo V, Israel G, King BS, Cohn S, Efron A, Pacheco AG, Moulton LH, Chaisson RE, Golub JE. The implementation of isoniazid preventive therapy in HIV clinics: the experience from the TB/HIV in Rio (THRio) study. AIDS. 2010 Nov;24 Suppl 5(Suppl 5):S49-56. doi: 10.1097/01.aids.0000391022.95412.a6. PMID 21079428
- [Background] Williams AB, Amico KR, Bova C, Womack JA. A proposal for quality standards for measuring medication adherence in research. AIDS Behav. 2013 Jan;17(1):284-97. doi: 10.1007/s10461-012-0172-7. PMID 22407465
- [Background] Marcellin F, Spire B, Carrieri MP, Roux P. Assessing adherence to antiretroviral therapy in randomized HIV clinical trials: a review of currently used methods. Expert Rev Anti Infect Ther. 2013 Mar;11(3):239-50. doi: 10.1586/eri.13.8. PMID 23458765
- [Background] Simoni JM, Huh D, Wang Y, Wilson IB, Reynolds NR, Remien RH, Goggin K, Gross R, Rosen MI, Schneiderman N, Arnsten J, Golin CE, Erlen JA, Bangsberg DR, Liu H. The validity of self-reported medication adherence as an outcome in clinical trials of adherence-promotion interventions: Findings from the MACH14 study. AIDS Behav. 2014 Dec;18(12):2285-90. doi: 10.1007/s10461-014-0905-x. PMID 25280447
- [Background] Kagee A, Nel A. Assessing the association between self-report items for HIV pill adherence and biological measures. AIDS Care. 2012;24(11):1448-52. doi: 10.1080/09540121.2012.687816. Epub 2012 Jun 7. PMID 22670758
- [Background] Marrazzo JM, Ramjee G, Richardson BA, Gomez K, Mgodi N, Nair G, Palanee T, Nakabiito C, van der Straten A, Noguchi L, Hendrix CW, Dai JY, Ganesh S, Mkhize B, Taljaard M, Parikh UM, Piper J, Masse B, Grossman C, Rooney J, Schwartz JL, Watts H, Marzinke MA, Hillier SL, McGowan IM, Chirenje ZM; VOICE Study Team. Tenofovir-based preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2015 Feb 5;372(6):509-18. doi: 10.1056/NEJMoa1402269. PMID 25651245
- [Background] Gandhi M, Ameli N, Bacchetti P, Anastos K, Gange SJ, Minkoff H, Young M, Milam J, Cohen MH, Sharp GB, Huang Y, Greenblatt RM. Atazanavir concentration in hair is the strongest predictor of outcomes on antiretroviral therapy. Clin Infect Dis. 2011 May;52(10):1267-75. doi: 10.1093/cid/cir131. PMID 21507924
- [Background] Gandhi M, Ameli N, Bacchetti P, Gange SJ, Anastos K, Levine A, Hyman CL, Cohen M, Young M, Huang Y, Greenblatt RM; Women's Interagency HIV Study (WIHS). Protease inhibitor levels in hair strongly predict virologic response to treatment. AIDS. 2009 Feb 20;23(4):471-8. doi: 10.1097/QAD.0b013e328325a4a9. PMID 19165084
- [Background] Gandhi M, Greenblatt RM. Hair it is: the long and short of monitoring antiretroviral treatment. Ann Intern Med. 2002 Oct 15;137(8):696-7. doi: 10.7326/0003-4819-137-8-200210150-00016. No abstract available. PMID 12379072
- [Background] Podsadecki TJ, Vrijens BC, Tousset EP, Rode RA, Hanna GJ. "White coat compliance" limits the reliability of therapeutic drug monitoring in HIV-1-infected patients. HIV Clin Trials. 2008 Jul-Aug;9(4):238-46. doi: 10.1310/hct0904-238. PMID 18753118
- [Background] Beumer JH, Bosman IJ, Maes RA. Hair as a biological specimen for therapeutic drug monitoring. Int J Clin Pract. 2001 Jul-Aug;55(6):353-7. PMID 11501221
- [Background] Liu AY, Yang Q, Huang Y, Bacchetti P, Anderson PL, Jin C, Goggin K, Stojanovski K, Grant R, Buchbinder SP, Greenblatt RM, Gandhi M. Strong relationship between oral dose and tenofovir hair levels in a randomized trial: hair as a potential adherence measure for pre-exposure prophylaxis (PrEP). PLoS One. 2014 Jan 8;9(1):e83736. doi: 10.1371/journal.pone.0083736. eCollection 2014. PMID 24421901
- [Background] van Zyl GU, van Mens TE, McIlleron H, Zeier M, Nachega JB, Decloedt E, Malavazzi C, Smith P, Huang Y, van der Merwe L, Gandhi M, Maartens G. Low lopinavir plasma or hair concentrations explain second-line protease inhibitor failures in a resource-limited setting. J Acquir Immune Defic Syndr. 2011 Apr;56(4):333-9. doi: 10.1097/QAI.0b013e31820dc0cc. PMID 21239995
- [Background] Baxi SM, Greenblatt RM, Bacchetti P, Jin C, French AL, Keller MJ, Augenbraun MH, Gange SJ, Liu C, Mack WJ, Gandhi M; Women's Interagency HIV Study (WIHS). Nevirapine Concentration in Hair Samples Is a Strong Predictor of Virologic Suppression in a Prospective Cohort of HIV-Infected Patients. PLoS One. 2015 Jun 8;10(6):e0129100. doi: 10.1371/journal.pone.0129100. eCollection 2015. PMID 26053176
- [Background] Koss CA, Natureeba P, Mwesigwa J, Cohan D, Nzarubara B, Bacchetti P, Horng H, Clark TD, Plenty A, Ruel TD, Achan J, Charlebois ED, Kamya MR, Havlir DV, Gandhi M. Hair concentrations of antiretrovirals predict viral suppression in HIV-infected pregnant and breastfeeding Ugandan women. AIDS. 2015 Apr 24;29(7):825-30. doi: 10.1097/QAD.0000000000000619. PMID 25985404
- [Background] Prasitsuebsai W, Kerr SJ, Truong KH, Ananworanich J, Do VC, Nguyen LV, Kurniati N, Kosalaraksa P, Sudjaritruk T, Chokephaibulkit K, Thammajaruk N, Singtoroj T, Teeraananchai S, Horng H, Bacchetti P, Gandhi M, Sohn AH. Using Lopinavir Concentrations in Hair Samples to Assess Treatment Outcomes on Second-Line Regimens Among Asian Children. AIDS Res Hum Retroviruses. 2015 Oct;31(10):1009-14. doi: 10.1089/AID.2015.0111. Epub 2015 Aug 26. PMID 26200586
- [Background] Huang Y, Gandhi M, Greenblatt RM, Gee W, Lin ET, Messenkoff N. Sensitive analysis of anti-HIV drugs, efavirenz, lopinavir and ritonavir, in human hair by liquid chromatography coupled with tandem mass spectrometry. Rapid Commun Mass Spectrom. 2008 Nov;22(21):3401-9. doi: 10.1002/rcm.3750. PMID 18837069
- [Background] Huang Y, Yang Q, Yoon K, Lei Y, Shi R, Gee W, Lin ET, Greenblatt RM, Gandhi M. Microanalysis of the antiretroviral nevirapine in human hair from HIV-infected patients by liquid chromatography-tandem mass spectrometry. Anal Bioanal Chem. 2011 Oct;401(6):1923-33. doi: 10.1007/s00216-011-5278-7. Epub 2011 Aug 17. PMID 21847531
- [Background] Hickey MD, Salmen CR, Tessler RA, Omollo D, Bacchetti P, Magerenge R, Mattah B, Salmen MR, Zoughbie D, Fiorella KJ, Geng E, Njoroge B, Jin C, Huang Y, Bukusi EA, Cohen CR, Gandhi M. Antiretroviral concentrations in small hair samples as a feasible marker of adherence in rural Kenya. J Acquir Immune Defic Syndr. 2014 Jul 1;66(3):311-5. doi: 10.1097/QAI.0000000000000154. PMID 24694932
- [Background] Gandhi M, Mwesigwa J, Aweeka F, Plenty A, Charlebois E, Ruel TD, Huang Y, Clark T, Ades V, Natureeba P, Luwedde FA, Achan J, Kamya MR, Havlir DV, Cohan D; Prevention of Malaria and HIV disease in Tororo (PROMOTE) study. Hair and plasma data show that lopinavir, ritonavir, and efavirenz all transfer from mother to infant in utero, but only efavirenz transfers via breastfeeding. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):578-84. doi: 10.1097/QAI.0b013e31829c48ad. PMID 24135775
- [Background] Baxi SM, Liu A, Bacchetti P, Mutua G, Sanders EJ, Kibengo FM, Haberer JE, Rooney J, Hendrix CW, Anderson PL, Huang Y, Priddy F, Gandhi M. Comparing the novel method of assessing PrEP adherence/exposure using hair samples to other pharmacologic and traditional measures. J Acquir Immune Defic Syndr. 2015 Jan 1;68(1):13-20. doi: 10.1097/QAI.0000000000000386. PMID 25296098
- [Background] Cohan D, Natureeba P, Koss CA, Plenty A, Luwedde F, Mwesigwa J, Ades V, Charlebois ED, Gandhi M, Clark TD, Nzarubara B, Achan J, Ruel T, Kamya MR, Havlir DV. Efficacy and safety of lopinavir/ritonavir versus efavirenz-based antiretroviral therapy in HIV-infected pregnant Ugandan women. AIDS. 2015 Jan 14;29(2):183-91. doi: 10.1097/QAD.0000000000000531. PMID 25426808
- [Background] Hahn JA, Emenyonu NI, Fatch R, Muyindike WR, Kekiibina A, Carrico AW, Woolf-King S, Shiboski S. Declining and rebounding unhealthy alcohol consumption during the first year of HIV care in rural Uganda, using phosphatidylethanol to augment self-report. Addiction. 2016 Feb;111(2):272-9. doi: 10.1111/add.13173. Epub 2015 Nov 5. PMID 26381193
- [Background] Geijo MP, Herranz CR, Vano D, Garcia AJ, Garcia M, Dimas JF. [Short-course isoniazid and rifampin compared with isoniazid for latent tuberculosis infection: a randomized clinical trial]. Enferm Infecc Microbiol Clin. 2007 May;25(5):300-4. doi: 10.1157/13102264. Spanish. PMID 17504682
- [Background] Sharma SK, Sharma A, Kadhiravan T, Tharyan P. Rifamycins (rifampicin, rifabutin and rifapentine) compared to isoniazid for preventing tuberculosis in HIV-negative people at risk of active TB. Cochrane Database Syst Rev. 2013 Jul 5;2013(7):CD007545. doi: 10.1002/14651858.CD007545.pub2. PMID 23828580
- [Background] Johnson JL, Okwera A, Hom DL, Mayanja H, Mutuluuza Kityo C, Nsubuga P, Nakibali JG, Loughlin AM, Yun H, Mugyenyi PN, Vernon A, Mugerwa RD, Ellner JJ, Whalen CC; Uganda-Case Western Reserve University Research Collaboration. Duration of efficacy of treatment of latent tuberculosis infection in HIV-infected adults. AIDS. 2001 Nov 9;15(16):2137-47. doi: 10.1097/00002030-200111090-00009. PMID 11684933
- [Background] Keeler E. Decision analysis. JAMA. 1977 May 30;237(22):2380. No abstract available. PMID 404441
- [Background] Gupta S, Abimbola T, Date A, Suthar AB, Bennett R, Sangrujee N, Granich R. Cost-effectiveness of the Three I's for HIV/TB and ART to prevent TB among people living with HIV. Int J Tuberc Lung Dis. 2014 Oct;18(10):1159-65. doi: 10.5588/ijtld.13.0571. PMID 25216828
- [Background] Pho MT, Swaminathan S, Kumarasamy N, Losina E, Ponnuraja C, Uhler LM, Scott CA, Mayer KH, Freedberg KA, Walensky RP. The cost-effectiveness of tuberculosis preventive therapy for HIV-infected individuals in southern India: a trial-based analysis. PLoS One. 2012;7(4):e36001. doi: 10.1371/journal.pone.0036001. Epub 2012 Apr 30. PMID 22558301
- [Background] Smith T, Samandari T, Abimbola T, Marston B, Sangrujee N. Implementation and Operational Research: Cost-Effectiveness of Antiretroviral Therapy and Isoniazid Prophylaxis to Reduce Tuberculosis and Death in People Living With HIV in Botswana. J Acquir Immune Defic Syndr. 2015 Nov 1;70(3):e84-93. doi: 10.1097/QAI.0000000000000783. PMID 26258564
- [Background] Hahn JA, Fatch R, Kabami J, Mayanja B, Emenyonu NI, Martin J, Bangsberg DR. Self-Report of Alcohol Use Increases When Specimens for Alcohol Biomarkers Are Collected in Persons With HIV in Uganda. J Acquir Immune Defic Syndr. 2012 Dec 1;61(4):e63-4. doi: 10.1097/QAI.0b013e318267c0f1. No abstract available. PMID 23138732
- [Background] Getahun H, Matteelli A, Abubakar I, Aziz MA, Baddeley A, Barreira D, Den Boon S, Borroto Gutierrez SM, Bruchfeld J, Burhan E, Cavalcante S, Cedillos R, Chaisson R, Chee CB, Chesire L, Corbett E, Dara M, Denholm J, de Vries G, Falzon D, Ford N, Gale-Rowe M, Gilpin C, Girardi E, Go UY, Govindasamy D, D Grant A, Grzemska M, Harris R, Horsburgh CR Jr, Ismayilov A, Jaramillo E, Kik S, Kranzer K, Lienhardt C, LoBue P, Lonnroth K, Marks G, Menzies D, Migliori GB, Mosca D, Mukadi YD, Mwinga A, Nelson L, Nishikiori N, Oordt-Speets A, Rangaka MX, Reis A, Rotz L, Sandgren A, Sane Schepisi M, Schunemann HJ, Sharma SK, Sotgiu G, Stagg HR, Sterling TR, Tayeb T, Uplekar M, van der Werf MJ, Vandevelde W, van Kessel F, van't Hoog A, Varma JK, Vezhnina N, Voniatis C, Vonk Noordegraaf-Schouten M, Weil D, Weyer K, Wilkinson RJ, Yoshiyama T, Zellweger JP, Raviglione M. Management of latent Mycobacterium tuberculosis infection: WHO guidelines for low tuberculosis burden countries. Eur Respir J. 2015 Dec;46(6):1563-76. doi: 10.1183/13993003.01245-2015. Epub 2015 Sep 24. PMID 26405286
- [Background] Gupta RK, Lucas SB, Fielding KL, Lawn SD. Prevalence of tuberculosis in post-mortem studies of HIV-infected adults and children in resource-limited settings: a systematic review and meta-analysis. AIDS. 2015 Sep 24;29(15):1987-2002. doi: 10.1097/QAD.0000000000000802. PMID 26266773
- [Background] Eby J, Chapman J, Marukutira T, Anabwani G, Tshume O, Lepodisi O, Dipotso T, Mokete K, Gross R, Lowenthal E. The adherence-outcome relationship is not altered by diary-driven adjustments of microelectronic monitor data. Pharmacoepidemiol Drug Saf. 2015 Dec;24(12):1313-20. doi: 10.1002/pds.3887. Epub 2015 Oct 12. PMID 26456482
- [Background] Berg KM, Arnsten JH. Practical and conceptual challenges in measuring antiretroviral adherence. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1(Suppl 1):S79-87. doi: 10.1097/01.qai.0000248337.97814.66. PMID 17133207
- [Background] Winhusen TM, Kropp F, Lindblad R, Douaihy A, Haynes L, Hodgkins C, Chartier K, Kampman KM, Sharma G, Lewis DF, VanVeldhuisen P, Theobald J, May J, Brigham GS. Multisite, randomized, double-blind, placebo-controlled pilot clinical trial to evaluate the efficacy of buspirone as a relapse-prevention treatment for cocaine dependence. J Clin Psychiatry. 2014 Jul;75(7):757-64. doi: 10.4088/JCP.13m08862. PMID 24911028
- [Background] Amico KR, Fisher WA, Cornman DH, Shuper PA, Redding CG, Konkle-Parker DJ, Barta W, Fisher JD. Visual analog scale of ART adherence: association with 3-day self-report and adherence barriers. J Acquir Immune Defic Syndr. 2006 Aug 1;42(4):455-9. doi: 10.1097/01.qai.0000225020.73760.c2. PMID 16810111
- [Background] Feldman BJ, Fredericksen RJ, Crane PK, Safren SA, Mugavero MJ, Willig JH, Simoni JM, Wilson IB, Saag MS, Kitahata MM, Crane HM. Evaluation of the single-item self-rating adherence scale for use in routine clinical care of people living with HIV. AIDS Behav. 2013 Jan;17(1):307-18. doi: 10.1007/s10461-012-0326-7. PMID 23108721
- [Background] Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav. 2008 Jan;12(1):86-94. doi: 10.1007/s10461-007-9261-4. Epub 2007 Jun 19. PMID 17577653
- [Background] Reid MC, Fiellin DA, O'Connor PG. Hazardous and harmful alcohol consumption in primary care. Arch Intern Med. 1999 Aug 9-23;159(15):1681-9. doi: 10.1001/archinte.159.15.1681. PMID 10448769
- [Background] McGinnis KA, Justice AC, Kraemer KL, Saitz R, Bryant KJ, Fiellin DA. Comparing alcohol screening measures among HIV-infected and -uninfected men. Alcohol Clin Exp Res. 2013 Mar;37(3):435-42. doi: 10.1111/j.1530-0277.2012.01937.x. Epub 2012 Oct 10. PMID 23050632
- [Background] Dhalla S, Kopec JA. The CAGE questionnaire for alcohol misuse: a review of reliability and validity studies. Clin Invest Med. 2007;30(1):33-41. doi: 10.25011/cim.v30i1.447. PMID 17716538
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Helander A, Hansson T. [National harmonization of the alcohol biomarker PEth]. Lakartidningen. 2013 Sep 25-Oct 8;110(39-40):1747-8. No abstract available. Swedish. PMID 24245431
- [Background] Wurst FM, Thon N, Yegles M, Schruck A, Preuss UW, Weinmann W. Ethanol metabolites: their role in the assessment of alcohol intake. Alcohol Clin Exp Res. 2015 Nov;39(11):2060-72. doi: 10.1111/acer.12851. Epub 2015 Sep 7. PMID 26344403
- [Background] Deschamps AE, Van Wijngaerden E, Denhaerynck K, De Geest S, Vandamme AM. Use of electronic monitoring induces a 40-day intervention effect in HIV patients. J Acquir Immune Defic Syndr. 2006 Oct 1;43(2):247-8. doi: 10.1097/01.qai.0000246034.86135.89. No abstract available. PMID 17003672
- [Background] Maruotti A. A two-part mixed-effects pattern-mixture model to handle zero-inflation and incompleteness in a longitudinal setting. Biom J. 2011 Sep;53(5):716-34. doi: 10.1002/bimj.201000190. Epub 2011 Aug 24. PMID 21887792
- [Background] Oni T, Burke R, Tsekela R, Bangani N, Seldon R, Gideon HP, Wood K, Wilkinson KA, Ottenhoff TH, Wilkinson RJ. High prevalence of subclinical tuberculosis in HIV-1-infected persons without advanced immunodeficiency: implications for TB screening. Thorax. 2011 Aug;66(8):669-73. doi: 10.1136/thx.2011.160168. Epub 2011 May 31. PMID 21632522
- [Background] Cox JA, Lukande RL, Nelson AM, Mayanja-Kizza H, Colebunders R, Van Marck E, Manabe YC. An autopsy study describing causes of death and comparing clinico-pathological findings among hospitalized patients in Kampala, Uganda. PLoS One. 2012;7(3):e33685. doi: 10.1371/journal.pone.0033685. Epub 2012 Mar 14. PMID 22432042
- [Background] Hoffmann CJ, Charalambous S, Thio CL, Martin DJ, Pemba L, Fielding KL, Churchyard GJ, Chaisson RE, Grant AD. Hepatotoxicity in an African antiretroviral therapy cohort: the effect of tuberculosis and hepatitis B. AIDS. 2007 Jun 19;21(10):1301-8. doi: 10.1097/QAD.0b013e32814e6b08. PMID 17545706
- [Background] Guo N, Marra CA, Marra F, Moadebi S, Elwood RK, Fitzgerald JM. Health state utilities in latent and active tuberculosis. Value Health. 2008 Dec;11(7):1154-61. doi: 10.1111/j.1524-4733.2008.00355.x. Epub 2008 May 16. PMID 18489493
- [Background] Kirenga BJ, Worodria W, Massinga-Loembe M, Nalwoga T, Manabe YC, Kestens L, Colebunders R, Mayanja-Kizza H. Tuberculin skin test conversion among HIV patients on antiretroviral therapy in Uganda. Int J Tuberc Lung Dis. 2013 Mar;17(3):336-41. doi: 10.5588/ijtld.12.0298. PMID 23407223
- [Background] Swaminathan S, Ramachandran R, Baskaran G, Paramasivan CN, Ramanathan U, Venkatesan P, Prabhakar R, Datta M. Risk of development of tuberculosis in HIV-infected patients. Int J Tuberc Lung Dis. 2000 Sep;4(9):839-44. PMID 10985652
- [Background] Whalen CC, Johnson JL, Okwera A, Hom DL, Huebner R, Mugyenyi P, Mugerwa RD, Ellner JJ. A trial of three regimens to prevent tuberculosis in Ugandan adults infected with the human immunodeficiency virus. Uganda-Case Western Reserve University Research Collaboration. N Engl J Med. 1997 Sep 18;337(12):801-8. doi: 10.1056/NEJM199709183371201. PMID 9295239
- [Background] Fitzgerald DW, Desvarieux M, Severe P, Joseph P, Johnson WD Jr, Pape JW. Effect of post-treatment isoniazid on prevention of recurrent tuberculosis in HIV-1-infected individuals: a randomised trial. Lancet. 2000 Oct 28;356(9240):1470-4. doi: 10.1016/S0140-6736(00)02870-1. PMID 11081529
- [Background] Golub JE, Cohn S, Saraceni V, Cavalcante SC, Pacheco AG, Moulton LH, Durovni B, Chaisson RE. Long-term protection from isoniazid preventive therapy for tuberculosis in HIV-infected patients in a medium-burden tuberculosis setting: the TB/HIV in Rio (THRio) study. Clin Infect Dis. 2015 Feb 15;60(4):639-45. doi: 10.1093/cid/ciu849. Epub 2014 Nov 2. PMID 25365974
- [Background] International Union Against Tuberculosis Committee on Prophylaxis. Efficacy of various durations of isoniazid preventive therapy for tuberculosis: five years of follow-up in the IUAT trial. International Union Against Tuberculosis Committee on Prophylaxis. Bull World Health Organ. 1982;60(4):555-64. PMID 6754120
- [Background] Nakagawa F, May M, Phillips A. Life expectancy living with HIV: recent estimates and future implications. Curr Opin Infect Dis. 2013 Feb;26(1):17-25. doi: 10.1097/QCO.0b013e32835ba6b1. PMID 23221765
- [Background] Mills EJ, Bakanda C, Birungi J, Mwesigwa R, Chan K, Ford N, Hogg RS, Cooper C. Mortality by baseline CD4 cell count among HIV patients initiating antiretroviral therapy: evidence from a large cohort in Uganda. AIDS. 2011 Mar 27;25(6):851-5. doi: 10.1097/QAD.0b013e32834564e9. PMID 21330903
- [Background] Lewden C, Chene G, Morlat P, Raffi F, Dupon M, Dellamonica P, Pellegrin JL, Katlama C, Dabis F, Leport C; Agence Nationale de Recherches sur le Sida et les Hepatites Virales (ANRS) CO8 APROCO-COPILOTE Study Group; Agence Nationale de Recherches sur le Sida et les Hepatites Virales (ANRS) CO3 AQUITAINE Study Group. HIV-infected adults with a CD4 cell count greater than 500 cells/mm3 on long-term combination antiretroviral therapy reach same mortality rates as the general population. J Acquir Immune Defic Syndr. 2007 Sep 1;46(1):72-7. doi: 10.1097/QAI.0b013e318134257a. PMID 17621240
- [Background] Badri M, Lawn SD, Wood R. Short-term risk of AIDS or death in people infected with HIV-1 before antiretroviral therapy in South Africa: a longitudinal study. Lancet. 2006 Oct 7;368(9543):1254-9. doi: 10.1016/S0140-6736(06)69117-4. PMID 17027731
- [Background] Masiira B, Baisley K, Mayanja BN, Kazooba P, Maher D, Kaleebu P. Mortality and its predictors among antiretroviral therapy naive HIV-infected individuals with CD4 cell count >/=350 cells/mm(3) compared to the general population: data from a population-based prospective HIV cohort in Uganda. Glob Health Action. 2014 Jan 15;7:21843. doi: 10.3402/gha.v7.21843. eCollection 2014. PMID 24433941
- [Background] Bendavid E, Grant P, Talbot A, Owens DK, Zolopa A. Cost-effectiveness of antiretroviral regimens in the World Health Organization's treatment guidelines: a South African analysis. AIDS. 2011 Jan 14;25(2):211-20. doi: 10.1097/QAD.0b013e328340fdf8. PMID 21124202
- [Background] Jelsma J, Maclean E, Hughes J, Tinise X, Darder M. An investigation into the health-related quality of life of individuals living with HIV who are receiving HAART. AIDS Care. 2005 Jul;17(5):579-88. doi: 10.1080/09540120412331319714. PMID 16036244
- [Background] Friend-du Preez N, Peltzer K. HIV symptoms and health-related quality of life prior to initiation of HAART in a sample of HIV-positive South Africans. AIDS Behav. 2010 Dec;14(6):1437-47. doi: 10.1007/s10461-009-9566-6. Epub 2009 May 13. PMID 19437112
- [Background] Shea KM, Kammerer JS, Winston CA, Navin TR, Horsburgh CR Jr. Estimated rate of reactivation of latent tuberculosis infection in the United States, overall and by population subgroup. Am J Epidemiol. 2014 Jan 15;179(2):216-25. doi: 10.1093/aje/kwt246. Epub 2013 Oct 18. PMID 24142915
- [Background] Durovni B, Saraceni V, Moulton LH, Pacheco AG, Cavalcante SC, King BS, Cohn S, Efron A, Chaisson RE, Golub JE. Effect of improved tuberculosis screening and isoniazid preventive therapy on incidence of tuberculosis and death in patients with HIV in clinics in Rio de Janeiro, Brazil: a stepped wedge, cluster-randomised trial. Lancet Infect Dis. 2013 Oct;13(10):852-8. doi: 10.1016/S1473-3099(13)70187-7. Epub 2013 Aug 16. PMID 23954450
- [Background] Bounthavong M, Hsu DI, Okamoto MP. Cost-effectiveness analysis of linezolid vs. vancomycin in treating methicillin-resistant Staphylococcus aureus complicated skin and soft tissue infections using a decision analytic model. Int J Clin Pract. 2009 Mar;63(3):376-86. doi: 10.1111/j.1742-1241.2008.01958.x. PMID 19222624
- [Background] Frey HC, Patil SR. Identification and review of sensitivity analysis methods. Risk Anal. 2002 Jun;22(3):553-78. PMID 12088234
- [Derived] Muyindike WR, Fatch R, Cheng DM, Emenyonu NI, Forman L, Ngabirano C, Adong J, Linas B, Jacobson KR, Hahn JA. Unhealthy Alcohol Use Is Associated With Suboptimal Adherence to Isoniazid Preventive Therapy in Persons With HIV in Southwestern Uganda. J Acquir Immune Defic Syndr. 2022 Dec 15;91(5):460-468. doi: 10.1097/QAI.0000000000003082. PMID 36044285
- See also: How AIDS Changed Everything: 2014 Global Statistics. UNAIDS;2015. — http://reliefweb.int/report/world/how-aids-changed-everything-mdg6-15-years-15-lessons-hope-aids-response
- See also: Guidelines for intensified tuberculosis case-finding and isoniazid preventive therapy for people living with HIV in resource-constrained settings. — http://apps.who.int/iris/bitstream/10665/44472/1/9789241500708_eng.pdf
- See also: UNAIDS Country Report, Uganda. 2014 — http://www.unaids.org/en/regionscountries/countries/uganda
- See also: Global Status Report on Alcohol and Health. Geneva: World Health Organization;2014 — http://www.who.int/substance_abuse/publications/global_alcohol_report/en/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an HIV clinic from April 2017 through December 2019.
Groups:
- INH and Vitamin B6: This was a single arm trial with a recruitment goal of 200 participants who reported current (prior 3 months) alcohol use, and 100 prior year abstinence from alcohol use. All participants were given 300 mg INH daily by mouth for 6 months, and 25 mg pyridoxine (vitamin B-6) daily by mouth for 6 months.
Period: Overall Study
Arm/Group | INH and Vitamin B6
Started | 302
Completed 3 Month Visit | 295
Completed 6 Month Visit | 289
Completed (Completed study enrollment and initiated isoniazid (INH) course.) | 301
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: 1 of 302 persons originally enrolled in the study was found to be ineligible during their baseline interview. They were disenrolled immediately and are excluded from all analyses, leaving 301 participants for analysis.
Groups:
- INH and Vitamin B6: This was a single arm trial; participants were given 300 mg INH daily by mouth for 6 months, and 25 mg pyridoxine (vitamin B-6) daily by mouth for 6 months.
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 301
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 40 [33 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 147
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 301

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Participants Experiencing a Grade 3/4 Hepatotoxicity
Description: Safety will be assessed by the occurrence of a Grade 3/4 hepatotoxicity at any time during the assigned treatment period.
Time Frame: Hepatotoxicity occurring during the six month course (180 pills) of isoniazid (INH), which may be taken over a maximum of 9 months.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 301
percent | 8.3 [5.4 to 12.0]

2. Secondary Outcome: Number of Participants Who Discontinued Treatment
Description: Lack of tolerability will be defined as any isoniazid (INH) treatment discontinuation prior to completion of the prescribed course (6 months of INH taken over a maximum period of 9 months) due to side effects or alanine transaminase (ALT)/aspartate transaminase (AST) elevations.
Time Frame: Six month course (180 pills) of isoniazid (INH), which may be taken over a maximum of 9 months.
Measure: Count of Participants; unit: Participants
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 301
Participants | 32

3. Secondary Outcome: Percentage of Participants With Suboptimal INH Medication Adherence
Description: Suboptimal INH adherence was defined as <90% of days with at least 1 electronic medication management (EMM) pill cap opening in the previous 90 days, at 3- and 6-months.
Time Frame: Adherence will be measured over the 6 months on INH or until INH discontinuation (whichever is shorter)
Population: 279/301 participants completed at least 1 study visit at either 3 or 6 months while on INH and are included here. 275 participants were included at 3 months; 264 participants were included at 6 months.
Measure: Number; unit: percentage of participants
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 279
percentage of participants
  at 3 months: number analyzed (Participants) | 275
  at 3 months | 31.3
  at 6 months: number analyzed (Participants) | 264
  at 6 months | 43.9
Statistical Analysis 1: Comparison: INH and Vitamin B6; Test type: Superiority; p < 0.01, Regression, Logistic — global p-value for 3-category alcohol use variable in a multivariable generalized estimating equation logistic regression model of sub-optimal INH adherence; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.94 to 2.71] — OR for participants with moderate alcohol use in the prior 3 months, compared to those with no alcohol use in the prior 3 months
Statistical Analysis 2: Comparison: INH and Vitamin B6; Test type: Superiority; p < 0.01, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.62 to 4.76] — OR is for participants with unhealthy alcohol use in the prior 3 months, compared to those with no alcohol use in the prior 3 months

4. Secondary Outcome: Self-reported INH Medication Adherence: Number of Days Taking INH in the Past 30 Days
Description: Participants were asked "In the past 30 days, how many days in total have you not taken your pill?" and were presented with a visual analog scale (VAS) to indicate the percentage of INH taken in the past 30 days. We converted the VAS percentage into number of days out of 30 to match the first question. Our final self-report measure was the minimum number of the 2 self-reported measurements.
Time Frame: Self-reported INH medication adherence via VAS will be measured 3- and 6- months after starting INH
Population: 290 unique participants are included here. 285 individuals are included at 3 months; 268 individuals are included at 6 months. Participants with missed visits or who were not taking INH (ie. due to either a temporary pause due to the COVID lockdown in Uganda, or because they were discontinued) were excluded.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 290
days
  at 3 months: number analyzed (Participants) | 285
  at 3 months | 30 [28 to 30]
  at 6 months: number analyzed (Participants) | 268
  at 6 months | 30 [27 to 30]

5. Secondary Outcome: Self-reported INH Medication Adherence by the Self Rating Single Item (SRSI) Scale
Description: The Self Rating Single Item (SRSI) adherence scale asks participants to rate their ability to take their medications as prescribed over the past 30 days. Participants reporting INH use in the prior 30 days at the 3- or 6-month interview are included here, and reported their INH adherence in the prior 30 days as excellent, very good, good, fair, poor, or very poor.
Time Frame: Self-reported INH medication adherence via SRSI will be measured 3- and 6- months after starting INH
Population: 280 unique participants are included here. 279 individuals are included at 3 months; 260 individuals are included at 6 months. Participants who reported no INH use in the prior 30 days were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 280
Participants
  At 3 months: number analyzed (Participants) | 279
  At 3 months: Excellent | 160
  At 3 months: Very good | 79
  At 3 months: Good | 38
  At 3 months: Fair | 0
  At 3 months: Poor | 2
  At 3 months: Very poor | 0
  At 6 months: number analyzed (Participants) | 260
  At 6 months: Excellent | 124
  At 6 months: Very good | 90
  At 6 months: Good | 41
  At 6 months: Fair | 4
  At 6 months: Poor | 0
  At 6 months: Very poor | 1

6. Other Pre Specified Outcome: INH Concentration in Hair: (INH Pmol + Acetyl INH Pmol) Per mg of Hair
Description: INH concentration in hair (pmol/mg) will be measured at 3- and 6- months during INH therapy.
Time Frame: Measured at 3- and 6- months after INH initiation
Population: We had funding to analyze the first shipped batch of hair (n=161 total visits, representing 97 unique participants) for INH.
Measure: Median (Inter-Quartile Range); unit: pmol/mg
Arm/Group | INH and Vitamin B6
Number analyzed (Participants) | 97
pmol/mg
  at 3 months: number analyzed (Participants) | 96
  at 3 months | 36.0 [18.7 to 63.3]
  at 6 months: number analyzed (Participants) | 65
  at 6 months | 37.8 [13.7 to 60.4]

7. Other Pre Specified Outcome: Number of Participants With Alanine Transaminase (ALT) or Aspartate Transaminase (AST) Elevations at Study Screening
Description: Alanine transaminase (ALT) or aspartate transaminase (AST) elevations (>2x the upper limit of normal) at study screening
Time Frame: Study screening visit
Population: People who completed liver transaminase testing as part of the screening for this study.
Measure: Count of Participants; unit: Participants
Groups:
- Study Screening: People who were screened as part of this study.
Arm/Group | Study Screening
Number analyzed (Participants) | 1303
Participants | 80

8. Other Pre Specified Outcome: Number of Participants With Latent Tuberculosis at Study Screening.
Description: Latent tuberculosis assessed at screening via tuberculin skin testing (TST). A TST induration >=5mm was considered positive for latent tuberculosis.
Time Frame: Study screening visit
Population: People who completed tuberculin skin testing (TST) as part of the study screening. People who did not return for the TST reading within the required window of 48-72 hours are excluded here.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Screening
Number analyzed (Participants) | 1156
Participants | 308

ADVERSE EVENTS:
Time Frame: Data were collected over the course of study participation, for a maximum of 42 months.
Arm/Group | INH and Vitamin B6
All-Cause Mortality (participants affected / at risk) | 2/301
Serious Adverse Events (participants affected / at risk) | 11/301
Other Adverse Events (participants affected / at risk) | 88/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INH and Vitamin B6 (N=301)
Elevated AST or ALT (Hepatobiliary disorders) | 6 (6) — Grade 4 aspartate transaminase (AST) or alanine transaminase (ALT) elevation defined as AST or ALT >=10 times the upper limit of normal (ULN).
Accident (Injury, poisoning and procedural complications) | 2 (2) — Injury from accident, resulting in hospitalization
Death (General disorders) | 2 (2) — Death - cause unknown
Septicemia (Infections and infestations) | 1 (1) — Septicemia causing hospitalization
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1) — Low hemoglobin, likely caused by persistent vaginal bleeding. Hospitalization
High blood pressure (Cardiac disorders) | 1 (1) — High blood pressure. Hospitalization.
Hospitalization (General disorders) | 1 (1) — Hospitalization due to dizziness, loss of appetite, nausea, paresthesia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INH and Vitamin B6 (N=301)
Grade 3: AST or ALT elevation (Hepatobiliary disorders) | 18 (18) — Grade 3 aspartate transaminase (AST) or alanine transaminase (ALT) elevation defined as AST or ALT >=5 to < 10 times the upper limit of normal (ULN).
Grade 2: AST or ALT elevation (Hepatobiliary disorders) | 62 (71) — Grade 2 aspartate transaminase (AST) or alanine transaminase (ALT) elevation defined as AST or ALT >2 to < 5 times the upper limit of normal (ULN).
PPD hypersensitivity (Immune system disorders) | 3 (3) — Hypersensitivity reaction to the tuberculin purified protein derivative (PPD) test. The total number at risk includes all people who received the PPD test as part of study screening.
Paresthesias (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Dizziness (General disorders) | 2 (2)
Angioedema (Immune system disorders) | 1 (1)
Allergic conjuctivitis (Eye disorders) | 1 (1)
Shooting pains (Nervous system disorders) | 1 (1)
Visual changes (blurring) (General disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Poor appetite (General disorders) | 1 (1)
Physically assaulted (Injury, poisoning and procedural complications) | 1 (1) — Physically assaulted by partner (grade 2 injury).
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) — Road traffic accident (grade 2 injury)
Hypertension (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03302299/Prot_SAP_001.pdf